CLINICAL TRIAL: NCT07050875
Title: Clinical Investigation to Validate the Safety and Performance of the ABLE Exoskeleton Device for Individuals With Acquired Brain Injury in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: Centro Europeo de Neurociencias (CEN) (Unknown); Cefine Neurología (CEFINE) (Unknown); Fundación Step by Step (SBS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABLEexoABI; CIV-25-04-052374 (Other: AEMPS)
Record Dates: First submitted 2025-06-16; First posted 2025-07-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acquired Brain Injury (Including Stroke)
Keywords: Gait training; Wearable exoskeleton; Acquired Brain Injury; Lower-limb exoskeleton; Multicenter
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait training with exoskeleton (Experimental): Participants will undergo a 10-session gait training program with the exoskeleton, twice a week for up to 6 weeks. Each session will last 60 minutes.
  Interventions: Device: ABLE Exoskeleton

INTERVENTIONS:
Device: ABLE Exoskeleton — Participants will undergo a 10-session gait training program with the exoskeleton, twice a week for up to 6 weeks. Each session will last 60 minutes.

SUMMARY:
The primary objective of the study is to validate the safety and clinical performance of the ABLE Exoskeleton device in people with acquired brain injury during a 10-session gait training program in a clinical setting.

The secondary objective of the study focuses on obtaining preliminary data on the potential clinical and psychosocial benefits of the product.

DETAILED DESCRIPTION:
This is a pre-post, multicenter, quasi-experimental study with an estimated duration of 17 weeks. The study will be conducted at the Centro Europeo de Neurociencias (CEN), Cefine Neurología (CEFINE), and Fundación Step by Step Foundation, where a minimum of 15 participants (5 per center) are expected to be recruited within a period of 8 weeks.

After obtaining informed consent, through the Patient Information Sheet and the Informed Consent Form, the selection of the participants will be carried out to determine their inclusion in the study. Subjects who do not meet all the inclusion and exclusion criteria during the screening visit will be excluded from the study. At the latest, one week after the screening visit, the participants will undergo a baseline assessment without the medical device.

Participants will undergo a 10-session training program with the ABLE Exoskeleton device for a maximum duration of 6 weeks. Sessions will be conducted 2 times per week. Each session will last approximately 60 minutes. During the training period, session data will be taken to assess the safety and clinical performance of the device. At the latest, one week after the last training session, a post-training assessment will be performed. Finally, two weeks after the last training session, a follow-up assessment will be made to the participants via a telephone call to review any adverse events (AE) reported between the end of the training and the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* Diagnosed with acquired brain injury (ABI)
* Currently undergoing outpatient physical therapy treatment in one of the investigation sites
* Ability to give informed consent

Exclusion Criteria:

* Significant osteoporosis that may increase the risk of fracture
* Unresolved fractures in the pelvis or extremities, or history of fragility fractures in the lower extremities in the last 2 years
* Spinal instability (or spinal orthoses, unless authorized by a physician)
* Severe spasticity: Level 4 on the Modified Ashworth Scale
* Orthostatic hypotension. Inability to tolerate a minimum of 10 minutes standing
* Uncontrolled autonomic dysreflexia
* Medical instability
* Unstable cardiovascular system (CVS), hemodynamic instability, untreated hypertension (SBP>140, DBP>90 mmHg), unresolved deep venous thrombosis (DVT), uncontrolled autonomic dysreflexia
* Serious comorbidities, including any condition that a physician deems inappropriate for use of the ABLE Exoskeleton or to complete participation in the study
* Skin integrity problems on the contact surfaces of the device or that would prevent sitting
* Grade I or higher on EPUAP (European Pressure Ulcer Advisory Panel, 2019) on areas that will be in contact with the exoskeleton
* Colostomy
* Anthropometric measurements outside the values compatible with ABLE Exoskeleton. In particular, height not between 1.5-1.9 m, or weight over 100 kg
* Anatomical constraints (such as leg length differences, users unable to position themselves inside the device) that are incompatible with the device
* Restrictions in range of motion that prevent normal gait from being achieved or preventing the completion of a normal transition from sitting to standing or standing to sitting
* Heterotopic ossification
* Known pregnancy or breastfeeding
* Cognitive impairment that results in the inability to follow simple instructions, particularly psychological or cognitive problems that do not allow a participant to follow study procedures
* Requires assisted ventilation.
* Scoliosis >40-50º Cobb angle.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Number and type of device-related Adverse Events | From baseline to follow-up (up to 2 weeks after end of intervention)
  To assess safety, the number of Severe Adverse Events (SAE), Adverse Events (AE) and drop-outs due to the device will be assessed and reported.
Level of Assistance (LoA) to don/doff the device | Up to 6 weeks
  Level of Assistance (LoA) to don/doff the device will be measured in every session. The level of assistance will be measured using a 6-item scale, from Total assistance to Independence, with Independence being the best outcome possible. Different assistance levels are defined taking into account the degree of participation of both the participant and the therapist on performing the activity.
Time taken to don/doff the device | Up to 6 weeks
  The time taken to don/doff the device will be measured in every session. Time will be measured in minutes and seconds for each activity. Donning time will start from the moment the participant is ready to transfer into the device until all the straps and clips are correctly tightened. Doffing time will start from the moment the participant starts taking off the device until they have completely removed it.
Number of steps walked | Up to 6 weeks
  In each gait training session, the number of steps taken (step count) with the device will be automatically measured and registered by the device
Distance walked | Up to 6 weeks
  In each gait training session, the distance walked (in meters) with the device will be automatically measured and registered by the device
Time spent upright and time spent walking | Up to 6 weeks
  In each gait training session, the time spent upright (in minutes) and the time spent walking (in minutes) with the device will be automatically measured and registered by the device
Number of therapists assisting the session | Up to 6 weeks
  In each gait training session, the number of therapists assisting will be recorded
Level of Assistance (LoA) during training | Up to 6 weeks
  Four therapy activity tasks will be attempted every session by the participant. The therapist will record the level of assistance required to complete each task during the session, using a 6-item scale, from Total assistance to Independence, with Independence being the best outcome possible. The tasks are the following: sit-to-stand, walk 10 meters, turn 180 degrees, and stand-to-sit.

SECONDARY OUTCOMES:
Lower extremity muscle strenght | At baseline (day 0) and post-training (up to 7 weeks)
  The Daniels Muscle Testing scale will be used to measure the strength of muscles in the lower extremities. Scores range from 0 (absence of muscle activity) to 5 (normal muscle activity)
Functional Ambulation Category (FAC) | At baseline(day 0) and post-training (up to 7 weeks)
  The patient's walking ability is evaluated with the Functional Ambulation Category (FAC) scale. It has 6 categories, from 0 (patient who is not able to walk) to 5 (independent patient who does not need any help to walk)
10-Meter Walking Test (10MWT) | At baseline(day 0) and post-training (up to 7 weeks)
  The 10-Meter Walking Test (10MWT) test measures the time a person needs to walk 10 meters. This test will be performed in the pre-post evaluations without the device to assess the change in the walking function after the training.
6-Minute Walk Test (6MWT) | At baseline (day 0) and post-training (up to 7 weeks)
  The 6-Minute Walk Test (6MWT) measures the distance a person can walk in 6 minutes. This test will be assessed at baseline and at the end of the gait training program without the device to assess the change in the walking function after the training
Timed Up and Go (TUG) | At baseline (day 0) and post-training (up to 7 weeks)
  The Timed Up-and-Go Test (TUG) measures the time it takes a person to get up from a chair, walk 3 meters, turn around, and sit down again. This test will be performed in the pre-post evaluations without the device to assess the change in the walking function after the training.
Trunk Impairment Scale (TIS) | At baseline (day 0) and post-training (up to 7 weeks)
  The Trunk Impairment Scale (TIS) measures the motor impairment of the trunk through the evaluation of static and dynamic sitting balance as well as coordination of trunk movement. The total score ranges from 0 (minimal performance) to 23 (perfect performance).
Berg Balance Scale (BBS) | At baseline and post-training (up to 7 weeks)
  The Berg Balance Scale (BBS) is used to assess the patient's ability to safely stabilize while performing certain tasks. It consists of a list of 14 items.
  Each item is evaluated through an ordinal scale ranging from 0 (lowest level of functionality) to 4 (highest level of functionality).
Modified Ashworth Scale (MAS) | At selection, baseline and post-training (up to 7 weeks)
  The Modified Ashworth Scale (MAS) measures spasticity in patients with lesions to the central nervous system. The scale assigns a grade of spasticity from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension).
Location and level of pain | From baseline to post-training (up to 7 weeks)
  The location and level of pain using the numeric rating scale (NRS) will be assessed. Each value is scored on a 0 to 10 scale, where 0 represents no pain and 10 represents the worst pain imaginable.
Borg Rating of Perceived Exertion | From baseline to post-training (up to 7 weeks)
  The Borg Rating of Perceived Exertion (RPE) scale is used to measure a person's perception of their effort and exertion, breathlessness, and fatigue during physical activity. Scores range from 6 (no exertion at all) to 20 (maximal exertion).
Functional Independence Measure (FIM) | At baseline and post-training (up to 7 weeks)
  The Functional Independence Scale (FIM) is a widely used instrument to assess the patient's outcomes and progress in rehabilitation programs. It is an indicator of disability, which measures how much assistance the patient needs to perform activities of daily living . It includes 18 activities that are measured on a 7-level scale, with 1 being indicative of total assistance and 7 of complete independence.
Level of motivation | At post-training (up to 7 weeks from baseline)
  Participants' perceptions on the level of motivation generated by the program with the ABLE Exoskeleton will be evaluated by the completion of a self-report questionnaire using a 7-point Likert scale. This questionnaire has been designed by the researchers.
Self-perceived impact on general health status | At post-training (up to 7 weeks)
  Participants' perceptions of the impact on their general health will be evaluated by the completion of a self-report questionnaire on the perceived impact on general health. This questionnaire has been designed by the researchers and intends to identify to what extent participants feel that the ABLE Exoskeleton contributed to a change in their health. The questionnaire covers 7 categories (cardiovascular system, musculoskeletal pain, neuropathic pain, bladder and bowel, spasticity, and sleep quality) using a 7-point Likert scale to assess the change.
Psychosocial Impact of Assistive Devices Scale (PIADS) score | At post-training (up to 7 weeks)
  The Psychosocial Impact of Assistive Devices Scale (PIADS) is a 26-item, self-reported questionnaire that provides a measure of user perception and other psychological factors associated with assistive technology devices. Scores range from -78 (maximum negative impact) to +78 (maximum positive impact). It will be used to assess the effects of the ABLE Exoskeleton on functional independence, well-being, and quality of life of participants after the training program experience
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) score | At post-training (up to 7 weeks)
  The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) is a 12-item outcome measure that assesses user satisfaction with two components (Device and Services) using a 5-point scale ranging from 1 (not satisfied) to 5 (very satisfied). Only the 8 items referred to the device will be evaluated from participants and the whole 12 items from the therapists to measure user satisfaction with the ABLE Exoskeleton after the training program experience

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Cefine Neurología (CEFINE), Culleredo, A Coruña
  - Fundación Step by Step, L'Hospitalet de Llobregat, Barcelona
  - Centro Europeo de Neurociencias (CEN), Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No